CLINICAL TRIAL: NCT05293938
Title: Study Evaluating the Effectiveness of Obeticholic Acid on Hepatic Real-World Outcomes in Patients With Primary Biliary Cholangitis
Brief Title: A Real-World Data Study to Evaluate the Effectiveness of OCA on Hepatic Outcomes in PBC Patients
Acronym: HEROES-PBC
Status: Withdrawn | Type: Observational
Why Stopped: A fundamental protocol deviation on data capture left the database no longer fit for purpose.
Sponsor: Intercept Pharmaceuticals (Industry)
Collaborators: Global PBC Study Group (Unknown); Target RWE (Industry); Syneos Health (Other); UK PBC Study Group (Unknown)
Responsible Party: Sponsor
Other Study IDs: 747-404
Record Dates: First submitted 2022-03-04; First posted 2022-03-24 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Primary Biliary Cholangitis
Keywords: Primary Biliary Cholangitis; Primary Biliary Cirrhosis; PBC; Hepatic Impairment; Liver
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — obeticholic acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OCA Treatment Group: PBC patients with a history of UDCA failure who initiated OCA in the study window (01 Jun 2015 to 31 Dec 2021)
  Interventions: Drug: Obeticholic Acid 5 MG; Drug: Obeticholic Acid 10 MG
- Control Group: PBC patients with a history of UDCA failure who were eligible but were not treated with OCA (or off-label fibrates) in the study window (01 Jun 2015 to 31 Dec 2021)
  Interventions: Drug: Standard of Care: UDCA

INTERVENTIONS:
Drug: Obeticholic Acid 5 MG — once daily, oral administration
  Other Names: Ocaliva
  Groups: OCA Treatment Group
Drug: Obeticholic Acid 10 MG — once daily, oral administration
  Other Names: Ocaliva
  Groups: OCA Treatment Group
Drug: Standard of Care: UDCA — No study medication is provided by the sponsor or by the investigators. The decision to initiate, continue or discontinue UDCA, or to modify UDCA dosing, is entirely at the discretion of the treating physician as per their standard of care and is in no way influenced by the sponsor or participating institutions. UDCA utilization is recorded and included in the study record.
  Groups: Control Group

SUMMARY:
This is an observational, retrospective cohort study, using the UK PBC registry, comparing patients with primary biliary cholangitis (PBC) who failed ursodeoxycholic acid (UDCA) treatment and were treated with obeticholic acid (OCA) to patients with PBC who failed UDCA treatment and were not treated with second-line therapy. The study is designed to evaluate the effectiveness of OCA. All patients who meet diagnostic criteria for PBC in the database between 01 Jun 2015 and 31 Dec 2021 and who meet all eligibility criteria will be considered for this study.

ELIGIBILITY:
Key Inclusion Criteria:

1. Definite or probable PBC diagnosis
2. UDCA failure
3. Age ≥18 years at the index date
4. Evaluable data for at least 12 months before the index date (inclusive)

Key Exclusion Criteria:

1. History or presence of other concomitant liver diseases
2. Patients with laboratory values indicative of hepatic decompensation or significant hepatobiliary injury
3. History of liver transplant
4. Evidence of OCA, fenofibrate, or bezafibrate use
5. History or presence of hepatic decompensating events
6. Participation in a clinical trial for a PBC medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who meet diagnostic criteria in UK PBC registry between 01 Jun 2015 and 31 Dec 2021 and who meet the eligibility criteria will be considered for the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Time to the first occurrence of the composite endpoint of all-cause death, liver transplant, or hepatic decompensation. | Time from index date to first occurrence of the composite endpoint events, assessed up to 62 months.

OTHER OUTCOMES:
Time to the first occurrence of all-cause death | Time from index date to first occurrence of all-cause death, assessed up to 62 months.
Time to the first occurrence of liver transplant | Time from index date to first occurrence of liver transplant, assessed up to 62 months.
Time to first occurrence of hepatic decompensation | Time from index date to first occurrence of hospitalization for hepatic decompensation, assessed up to 62 months.

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Szczech, MD, Study Director — Intercept Pharmaceuticals
Locations (1):
- Intercept Pharmaceuticals, Inc, San Diego, California, United States